CLINICAL TRIAL: NCT01467869
Title: The Miami Project Male Fertility Program
Brief Title: Male Fertility Program
Acronym: MFP
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Emad Ibrahim, Instructor, University of Miami
Other Study IDs: 19910013
Record Dates: First submitted 2011-09-29; First posted 2011-11-09 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury
Keywords: abnormal semen; assisted conception
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Following spinal cord injury, most men are infertile and require medical assistance to father children. The conditions that contribute to their infertility are erectile dysfunction, ejaculatory dysfunction, and semen abnormalities. The Miami Project Male Fertility Program is a research study designed to understand and improve impairments to male fertility resulting from spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Any man with spinal cord injury over the age of 18. Control Subjects will be any healthy man over the age of 18 with no recent history of infertility

Exclusion Criteria:

* Women will be excluded.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Spinal cord injured men
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 1991-01 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
spinal cord injury (SCI) subjects will learn the best method to obtain their semen and of their possible options for assisted conception. | 2 visits; subjects will provide samples each month up to an average of 2-3 months
  Studies in the male fertility program will investigate the fertility potential of spinal cord injured men by retrieving semen which will be analyzed for sperm count, motility, morphology, etc., and correlated with patient variables such as age, time of injury, level of injury, bladder management, history of UTI's, hormonal status, etc. the outcome of the research will improve fertility in men with spinal cord injury.

CONTACTS AND LOCATIONS:
Overall Officials: Emad Ibrahim, MD, Principal Investigator — University of Miami
Locations (1):
- The Maimi Project to Cure Paralysis, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ibrahim E, Aballa TC, Lynne CM, Brackett NL. Oral probenecid improves sperm motility in men with spinal cord injury. J Spinal Cord Med. 2018 Sep;41(5):567-570. doi: 10.1080/10790268.2017.1320875. Epub 2017 May 2. PMID 28464732
- See also: Related Info — http://www.themiamiproject.org